CLINICAL TRIAL: NCT03184207
Title: A Systematic Ultrasound Assessment During Intubation Procedure to Predict Cardiovascular Collapse Related to Intubation in the Intensive Care Unit: a Prospective, Multiple-center Study
Brief Title: A Systematic Echography During Intubation Procedure to Predict Cardiovascular Collapse
Acronym: EPIC
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: EPIC ( 29BRC17.0047)
Record Dates: First submitted 2017-04-13; First posted 2017-06-12 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-07

CONDITIONS: Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the operating room, most intubation procedures (IP) are scheduled and performed on hemodynamically stable patients. In the ICU, IP is frequently performed in emergent patients, because of unstable hemodynamics and/or acute respiratory failure, and complicated by a subsequent cardiovascular collapse. Transthoracic echocardiography (TTE) has become readily available in most ICUs for several years. Echocardiography enables to perform a noninvasive hemodynamic evaluation (cardiac function and volemia status).

We hypothesized that performing a TTE prior to IP may help to predict cardiovascular collapse and its components.

ELIGIBILITY:
Inclusion Criteria:

Patient requiring endotracheal intubation

Exclusion Criteria:

* Age < 18 yrs
* Pregnancy
* Amputation of a lower limb
* Passing leg raising contraindication: intracranial hypertension with invasive monitoring, fracture of the pelvis or limbs
* Patients under administrative protective measures
* Severe cardiovascular collapse before intubation
* Severe cardiogenic pulmonary oedema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient admitted to ICU
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2017-06-21 (Actual); Study Completion 2018-10-19 (Actual)

PRIMARY OUTCOMES:
Subsequent cardiovascular collapse related to intubation | Within 15 minutes of intubation
  Mean arterial pressure drop < 60 mmHg

SECONDARY OUTCOMES:
Ultrasound parameters to predict fluid responsiveness | 30 minutes before intubation, less than 30 minutes after intubation, 1 minutes after lifting legs and 3 hours after intubation
  Transthoracic echocardiography parameters to predict fluid responsiveness

CONTACTS AND LOCATIONS:
Overall Officials: JEAN-MICHEL Vanessa, M.D., Principal Investigator — CHRU Brest Hospital Brittany Occidental University
Locations (3):
- France (3):
  - Hôpital d'Instruction des Armées Clermont Tonnerre, Brest
  - CHRU de Brest, Brest
  - Centre Hospitalier des Pays de Morlaix, Morlaix

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jaber S, Jung B, Corne P, Sebbane M, Muller L, Chanques G, Verzilli D, Jonquet O, Eledjam JJ, Lefrant JY. An intervention to decrease complications related to endotracheal intubation in the intensive care unit: a prospective, multiple-center study. Intensive Care Med. 2010 Feb;36(2):248-55. doi: 10.1007/s00134-009-1717-8. Epub 2009 Nov 17. PMID 19921148